CLINICAL TRIAL: NCT01545882
Title: A Phase II Study of Degarelix in the Management of Non-Metastatic Hormone-Refractory Prostate Cancer
Acronym: OTT10-06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative study; Principal Investigator chose to prematurely terminate the study.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-059; OTT10-06 (Other: The Ottawa Hospital Cancer Centre)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Prostatic Neoplasms
Keywords: prostate; hormone-resistant; degarelix; firmagon; anti-androgens; total androgen blockade; injection
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental): Degarelix treatment will consist of a starting dose of 240mg injected subcutaneously (s.c) and monthly s.c. maintenance doses of 80mg for a total duration of 6 months.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Treatment will consist of a starting dose of 240mg injected subcutaneously (s.c) and monthly s.c. maintenance doses of 80mg for a total duration of 6 months.
  Other Names: Firmagon

SUMMARY:
This study is being offered to patients who have hormone resistant prostate cancer (HRPC). This means that their prostate cancer is no longer responding to standard hormonal therapy.

The purpose of this study is to determine whether Degarelix will be able to stop the PSA from rising in patients with hormone resistant prostate cancer.

DETAILED DESCRIPTION:
This is a phase II study of a GnRH antagonist drug, Degarelix, for use in hormone resistant prostate cancer patients who have had biochemical PSA progression despite the use of total androgen blockade therapy. Patients will receive at least six monthly injections of Degarelix unless the patient shows radiographic or symptomatic disease progression, intolerable toxicity or decides to withdraw from the study. Patients will be evaluated for measures of efficacy, toxicity and disease progression during treatment and afterwards until radiologically confirmed metastatic disease progression or until the patient is removed from the study.

Overall objective:

The efficacy of Degarelix as a treatment for HRPC will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Prior trial of total androgen blockade
* Confirmed biochemical PSA progression on agonist therapy, defined as ≥ 50% increase in PSA between 2 measurements, taken at least 1 week apart. In patients that are currently on total androgen blockade (LHRH agonist plus non-steroidal anti-androgen) there must be a trial withdrawal of androgen receptor antagonists to ensure that there is no PSA response (6 weeks for bicalutamide and 4 weeks for flutamide or nilutamide).
* Radiologically confirmed non-metastatic disease within 90 days of registration based on negative chest radiographs, CT Scan Abdomen/Pelvis and Bone scan
* ECOG ≤ 2
* Age ≥ 18 years
* Serum testosterone of ≤ 50 mg/dl
* PSA ≥ 2.0 ng/ml
* White blood cell count ≥ 3000/mm3
* Platelets ≥ 100,000/mm3
* Serum creatinine ≤ 1.5 x upper limits of normal
* Bilirubin ≤ 1.5 x upper limits of normal
* Alanine transaminase ≤ 1.25 x upper limits of normal
* Estimated life expectancy of at least 12 months
* Able and willing to sign informed consent

Exclusion Criteria:

* Prior treatment with chemotherapy, radiopharmaceuticals, estrogen, PC-SPES, ketoconazole or other second line hormonal therapy (other than non-steroidal anti-androgens or Androcur)
* Known allergy to GnRH agonists or antagonists
* Previous treatment with Degarelix
* Major surgery within 4 weeks of registration
* Grade ≥ 3 peripheral neuropathy
* Severe, active co-morbidity such as unstable angina, congestive heart failure or myocardial infarction within the last 6 months or congenital long QT syndrome
* Acute deep vein thrombosis or pulmonary embolism
* Taking anti-arrhythmia medication
* Second malignancy other than non-melanoma skin cancer unless disease free ≥ 5 years.
* Prior orchiectomy for prostate cancer
* PSA > 100 ng/mL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
PSA Progression | Monthly for 6 months then every 3 months
  Blood work will be done once a month during the 6 months of treatment then every 3 months until disease progression or participant withdrawal

SECONDARY OUTCOMES:
Time to Disease progression | Monthly for 6 months then every 3 months
  Blood work will be done once a month during the 6 months of treatment then every 3 months until disease progression or participant withdrawal
The efficacy of Testosterone, LH and FSH suppression with Degarelix | Monthly for 6 months then every 3 months
  Blood work will be done once a month during the 6 months of treatment then every 3 months until disease progression or participant withdrawal
The impact of monthly injections of Degarelix on Health Related Quality of Life Issues in patients with prostate cancer | Month 3 and 6 then every 3 months
  The EPIC-26 Expanded Prostate Cancer Index Composite is used to measure quality of life issues in patients with prostate cancer. The questionnaire will be done months 3 and 6 then every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Malone, Dr., Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (3):
- Canada (3):
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margeret Hospital, Toronto, Ontario